CLINICAL TRIAL: NCT01397630
Title: Accelerate Versus Gradual Titration of Oxytocin Dose for Labour Dystocia: A Pilot Study
Brief Title: Accelerated Titration of Oxytocin for Nulliparous Patients With Labour Dystocia: ACTION Pilot Study
Acronym: ACTION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to budgetary concerns, the TSC decided it best to adjust sample size as there was sufficient data to assess feasibility. Recruitment was terminated early.
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); The Ottawa Hospital (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Sainte Justine Hospital Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-521
Record Dates: First submitted 2011-07-07; First posted 2011-07-19 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Labour Dystocia
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Accelerated Oxytocin Titration (Experimental)
  Interventions: Drug: Oxytocin
- Gradual Oxytocin Titration (Active Comparator)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Accelerated Oxytocin Titration
  Other Names: Pitocin, Syntocinon, Uteracon

SUMMARY:
The ultimate objective is to test the hypothesis that an 'accelerated titration' protocol for labour augmentation with oxytocin reduces the risk of caesarean births relative to a 'gradual titration' protocol.

The aims of this pilot feasibility are:

1. To assess the feasibility of a large multi-centre randomized control trial comparing the two above oxytocin protocols (accelerated titration versus gradual titration for correction of dystocia).
2. More specifically, to identify potential challenges in the study implementation, particularly with respect to patient recruitment, randomization, blinding, and compliance/adherence to the labour management guidelines and study protocols.
3. To obtain preliminary data on the acceptability of the accelerated oxytocin titration protocol among obstetrical providers and participants.

DETAILED DESCRIPTION:
There has been a steady increase in the rate of Caesarean births in Canada and worldwide. Almost half of all primary caesarean sections are performed for labour dystocia - when labour is abnormally slow or when there is no further progression in cervical dilatation. When dystocia occurs, oxytocin is used to increase the frequency and intensity of uterine contractions, with the goal of achieving full cervical dilatation and a vaginal birth. The actual dose required to produce a clinical response (progressive cervical dilatation) varies greatly from patient to patient. There is a wide range of oxytocin regimens currently in use. They may be broadly categorized as being of two types: 1) those involving a gradual titration of oxytocin dose (or 'low dose') and 2) those with accelerated oxytocin titration (also called 'high dose').

In fact, the frequently used terms 'low dose' and 'high dose' are to a certain extent misnomers. Both protocols titrate oxytocin dose to achieve the desired 'physiological frequency' of uterine contractions (usually 4 to 5 contractions in a 10 minute interval) that are normally sufficient to result in progressive labour. Thus, the target dose should, theoretically, be identical and independent of the rate of increase of oxytocin. These protocols differ mainly in the rate at which the desired physiologic response is achieved. While most patients achieve a response to stimulation at oxytocin concentrations between 4 and 10 mU per minute, a proportion of nulliparae require higher doses of oxytocin. Accelerated titration protocols are also frequently associated with a higher maximum concentration of oxytocin. While, most Canadian birthing centres currently follow a 'gradual titration' or 'low dose' protocol, there is evidence that 'accelerated titration' or 'high dose' protocols may be more effective in correcting dystocia and in preventing caesarean section. It is postulated that by more rapidly progressing to the required therapeutic dose, cervical dilatation is achieved more rapidly, the likelihood of a spontaneous vaginal birth is increased, and the risk of occurrence of complications resulting from prolonged labour (such as infection and maternal fatigue) is reduced.

ELIGIBILITY:
Inclusion Criteria:

1. Capability of participant to comprehend English and/or French and to comply with study requirements
2. ≥ 18 years of age at time of consent
3. Nulliparity
4. Singleton pregnancy
5. Cephalic Presentation
6. No contraindications to trial of labour or vaginal birth
7. Term pregnancy (37+0 to 42+0 weeks gestation)
8. Spontaneous onset of labour
9. In the ACTIVE phase of the FIRST stage of labour. Active labour is defined as:

   1. The presence of regular uterine contractions
   2. Cervical dilatation of ≥ 3 cm
   3. Cervical effacement of at least 80% (cervical length < 1cm)
10. DYSTOCIA in the ACTIVE phase of FIRST stage of labour established by the Physician.

    1. Cervical change of < 0.5 cm/hour over four hours OR
    2. NO cervical change in 2 hours
11. Ruptured amniotic membranes of at least 30 minutes
12. Normal fetal heart rate pattern at the time of randomization

Exclusion Criteria:

1. Serious medical condition (severe cardiac, pulmonary, or renal disease)
2. Known fetal anomaly
3. Known sensitivity to oxytocin
4. Contraindications to labour or vaginal birth (uterine scar)
5. Induced labour (using any method)
6. Oxytocin use prior to randomization
7. Second stage of labour
8. Suspected IUGR (<5th percentile)
9. Suspected macrosomia at term (>4500 grams)
10. Oligohydramnios (no 2x2 pocket of fluid on ultrasound prior to rupture of amniotic membranes)
11. Abnormal FHR pattern at the time of randomization
12. Suspected chorioamnionitis
13. Severe pre-eclampsia
14. Suspected placental abruption

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Consent Rate | From screening for eligibility until randomization (up to 5 weeks)
  1. The proportion of patients who are eligible and thus meet inclusion/exclusion criteria at time of labour onset
  2. The proportion of eligible participants who consent to participate and are randomized
Protocol Violation Rate | From admission to a hospital for delivery until delivery (up to 1 week)
  a) The proportion among those randomized of deviation from study protocol with regards to duration of oxytocin augmentation prior to operative intervention
Maternal satisfaction | from hospital admission to 4 weeks postpartum
  1. Pain score on visual analog scale during labour and delivery
  2. North Bristol modified Mackey childbirth satisfaction rating scale

SECONDARY OUTCOMES:
Caesarean section rate | From admission to a hospital for delivery until delivery (up to 1 week)
Rate of Maternal and Fetal/Neonatal Adverse Events | From admission to the hospital for delivery until discharge of the baby from the neonatal intensive care unit (up to 4 weeks after birth)
  1. Rate of tachysystole and hyperstimulation
  2. Rate of abnormal FHR pattern
  3. Composite index of adverse fetal outcome (cord arterial pH < 7.1, base deficit ≥ 12 mmol/L, 5 minute Apgar score ≤ 7)
  4. Admission of a term infant to the neonatal intensive care unit
  5. Proportion requiring unblinding of protocol

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Dy, MD, Principal Investigator — Ottawa Hospital Research Institute; Shu Qin Wei, MD, PhD, Principal Investigator — Sainte-Justine Hospital
Locations (2):
- Canada (2):
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sainte-Justine Hospital, Montreal, Quebec